CLINICAL TRIAL: NCT03262363
Title: Interaction of Polymorphism rs35652124 With Curcumin Supplementation on NFE2L2 Gene Expression, Antioxidant Capacity and Renal Function in Patients With Early Diabetic Nephropathy
Brief Title: Curcumin on NFE2L2 Gene Expression, Antioxidant Capacity and Renal Function According to rs35652124 in Diabetic Nephropathy
Acronym: CURCUNRF2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidad de Investigacion Medica en Enfermedades Renales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UIMER002
Record Dates: First submitted 2017-08-18; First posted 2017-08-25 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2017-09

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus, Type 2; Polymorphism
Keywords: nutrigenomics; Diet-gene interaction,; Curcumin,; Antioxidants,; Human NFE2L2 protein,; Polymorphism,; Diabetes,; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: The study starts from the classification of patients according to the genotype for the rs35652124 polymorphism (-653G>A) of the NFE2L2 gene. Two Experimental groups and two Control groups will be formed according to the following:
  Experimental group 1: Diabetic patients with early CKD homozygous for the -653G (G/G) allele of the NFE2L2 gene that will receive curcumin.
  Experimental group 2: Diabetic patients with early CKD carrying the allele -653A (G/A or A/A) of the NFE2L2 gene that will receive curcumin.
  Control group 1: Diabetic patients with early CKD homozygous for the -653G (G/G) allele of the NFE2L2 gene receiving placebo.
  Control group 2: Diabetic patients with early CKD carrying the allele -653A (G/A or A/A) of the NFE2L2 gene who will receive placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient Blinding: Patients with EDN will be blinded to the intervention they will receive Evaluator Blinding: The principal investigator will be blinded to the intervention that patients will receive (curcumin or placebo), but will know the genotype distribution in both Experimental and Placebo groups. The external investigator will be blinded to the knowledge of the patients genotype, but will know the intervention group to which each patient was assigned according to a registry (but will not know the identity of the patients). The Doctorate Program Student will be blinded to the distribution of patients genotype and the type of intervention patients will receive.
  Statistical Blinding: An associated researcher will be blinded to the distribution of patients genotype and the type of intervention patients will receive, but not to the knowledge of the database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin/NFE2L2 A>G (Experimental): Patients in Experimental group 1 and 2 will receive 800 mg/day of curcumin (for which a bioavailability of about 90% has been demonstrated and greater than other curcuminoids, administered in two doses of 400 mg each (the presentation will be in capsules containing 400 mg of THC).
  Interventions: Combination Product: Curcumin/NFE2L2 A>G
- Placebo/NFE2L2 A>G (Placebo Comparator): Patients in control group 1 and 2, the placebo intervention will consist of administering sucralose capsules (a substance lacking pharmacological action, with no active principle and a lower intake of glucose compared to sucrose). Patients will receive 300 mg/day of sucralose distributed in two doses of 150 mg each.
  Interventions: Combination Product: Placebo/NFE2L2 A>G

INTERVENTIONS:
Combination Product: Curcumin/NFE2L2 A>G — The administration will be orally and the patient will be instructed to take two capsules per day for one week, one in the morning 15 minutes before breakfast and another at night 15 minutes before dinner, accompanied by a cup of 240 mL of pure water. It will be indicated to continue with their usual medical treatment.
  Other Names: Curcumin group
  Arms: Curcumin/NFE2L2 A>G
Combination Product: Placebo/NFE2L2 A>G — The administration will be orally and the patient will be instructed to take two capsules for 24 weeks, one in the morning 15 minutes before breakfast and another in the evening 15 minutes before dinner, accompanied by a 240 mL cup of pure water. They will be advised to continue their usual medical treatment.
  Other Names: Placebo group
  Arms: Placebo/NFE2L2 A>G

SUMMARY:
The increase in the prevalence of diabetes mellitus (DM) is one of the greatest public health challenges worldwide. Epidemiological studies have shown that DM is the leading cause of chronic kidney disease (CKD) in patients initiating renal replacement therapy. In our country, diabetes accounts for about 60% of all incidents of dialysis. On the other hand, CKD is currently considered a noxious disease because patients not only have the likelihood of progression to end-stage renal disease (ESRD), but because these renal alterations are associated with an increased risk of cardiovascular complications and premature death for the same cause. Most studies have focused on traditional risk factors (poor diet, physical inactivity and obesity) for the development and progression of renal damage, and less information exists on non-traditional factors such as oxidative stress and mainly, the low antioxidant response that characterizes both DM and nephropathy. In addition, there is a great variation in the susceptibility to and progression of kidney disease between different populations that is not explained by the presence of traditional factors and that could be triggered by genetic variations and its interaction with other components related to the environment and lifestyle. Fortunately, there is sufficient scientific evidence that early detection and modification of negative lifestyle factors can not only delay or halt the progression of the renal function decline to ESRD but can also significantly reduce the incidence of cardiovascular disease leading to premature death in most of these patients. Therefore, it is suggested that this risk may be determined by the interaction of lifestyle factors with the presence of susceptibility alleles, which may vary from one population to another. It is now known that hyperglycemia causes a state of oxidative stress and inflammation that can be counteracted by diet supplementation with some natural antioxidants such as curcumin. It has been shown that this molecule has multiple pharmacological properties: antioxidant, anti-inflammatory, cardioprotective, renoprotective, among others. In clinical trials a positive effect of curcumin has been seen in the treatment of diabetes and its complications. This has generated a relative optimism in the search for new curcumin treatment targets where oxidative stress is of great relevance, as is the case with CKD. However, there are still doubts about its efficacy as an adjuvant in the prevention of CKD. Additionally, the role played by interindividual variability in genes involved in the mechanism of action of curcumin is still incipient, more studies in this knowledge area are necessary.

DETAILED DESCRIPTION:
Aim: To evaluate the interaction between rs35652124 polymorphism and curcumin supplementation on the levels of NFE2L2 gene expression, antioxidant capacity and renal function in patients with early diabetic nephropathy (EDN).

Subjects and Methods. Parallel clinical trial with randomized and triple blind. From a database of diabetic patients newly diagnosed with CKD, those with EDN will be identified and located by telephone to complete a total of 275 subjects over 18 years of age. Subsequently, they will be cited in the office of Biomedical Unit 02, will verify that they meet the selection criteria, will be informed about the objectives of the study and invited to participate. Those who agree to participate will be given an informed consent letter, they will be asked to read it carefully and if they have any doubts, they will be clarified at the moment. Once they have signed the written consent they will be cited for the first blood sample collecting (5 mL) to be used for genomic DNA extraction and genotyping for the rs35652124 polymorphism. All patients entering the study will undergo a physical and dietary examination and will record the data on a clinical record card. They will be prescribed a meal plan according to ADA recommendations and K/DOQI guidelines two weeks prior (week <2) at the start of the clinical trial, which will be maintained throughout the follow-up. They will then be scheduled monthly for medical and nutritional assessment. At the visits of weeks 2, 0 (start of supplementation), 12, and 24, three peripheral blood tubes (5 mL each) will be drawn. The first, to extract total mRNA and expression analysis of the NFE2L2 gene, the second, to determine the levels of NRF2, SOD, GPx and HO1 and the third, to perform renal function tests and control of possible confounding variables (creatinine, glucose, glycosylated hemoglobin, lipid profile and uric acid). In addition, they will be asked to collect a sample of the first morning urine to quantify albuminuria/creatinuria on the same day that blood samples were taken. The time of the study since the first evaluation is 26 weeks and the total number of medical and nutrition visits will be six, one monthly. Genotyping will be performed by polymerase chain reaction (PCR) coupled to four pairs of oligonucleotide primers specific for the alleles of interest. The gene expression assay will be performed by real-time PCR, while the determination of the concentrations of NRF2, SOD, GPx and HO1 will be carried out by the ELISA method with kits designed for this purpose. The analysis of the data includes descriptive statistics expressed in averages and standard or median deviations according to the parametric or non-parametric distribution, the nominal variables will be presented as numbers or percentages and the comparison between these will be by Chi square or Fisher exact. Inferential statistics included U-Mann Whitney or Student t tests for independent and paired samples as appropriate to evaluate the NRF2, SOD, GPx and HO1 concentrations with the different interventions and the individuals in the control group. A covariance analysis will be performed taking into consideration the factor supplementation, genetic factor and the interaction of both with the concentrations of NRF2. A value of p<0.05 and 95% CI will be considered significant.

Resources and infrastructure. The CIBO and the Medical Research Unit in Renal Diseases have the human resources to coordinate and develop the present research. Also, they have the necessary infrastructure and equipment to carry out the procedures contemplated in this project. The project will be submitted to calls for funding to obtain the necessary resources for its development.

ELIGIBILITY:
Inclusion Criteria:

* With T2DM according to the American Diabetes Association
* With any time of T2DM evolution
* With CKD stage 1-3a according to the K/DIGO guidelines

Exclusion Criteria:

* Incomplete evaluations
* That they have not been attached to the assigned intervention with an established frequency of <80%
* Decide to withdraw from the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline expression Gen NFE2L2 at 3 months | Baseline at 3 months
  mRNA and active protein NRF2
Change from Baseline expression Gen NFE2L2 at 6 months | Baseline at 6 months
  mRNA and active protein NRF2
Change from Antioxidant capacity at 3 months | Baseline at 3 months
  Superoxide dismutase, hemoxygenase 1, Glutathion peroxidase using the ELISA technique
Change from Antioxidant capacity at 6 months | Baseline at 6 months
  Superoxide dismutase, hemoxygenase 1, Glutathion peroxidase using the ELISA technique
Change from Renal Function at 3 months | Baseline at 3 months
  Glomerular Filtration Rate (Serum creatinine) and Albuminuria (Albumin/Creatinine Ratio)
Change from Renal Function at 6 months | Baseline at 6 months
  Glomerular Filtration Rate (Serum creatinine) and Albuminuria (Albumin/Creatinine Ratio)

CONTACTS AND LOCATIONS:
Locations (1):
- Umae Hospital de Especialidades, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] United States Renal Data Sytem. 2016 USRDS annual data report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases. Bethesda, MD, 2016.
- [Background] Gutiérrez JP, Rivera Dommarco J, Shamah Levy T, et al. Encuesta Nacional de Salud y Nutrición 2012. Resultados Nacionales. Cuernavaca, México: Salud Publica Mex; 2012.
- [Background] Hernández Ávila M, Gutiérrez JP, editores. Diabetes mellitus: la urgencia de reforzar la respuesta en políticas públicas para su prevención y control. Cuernavaca, México: Salud Publica Mex; 2012.
- [Background] Asociación Latinoamericana de Diabetes (ALAD). Guías ALAD sobre el diagnóstico, control y tratamiento de la diabetes mellitus Tipo 2 con medicina basada en evidencia. 1a ed. Latinoamérica: ALAD; 2013.
- [Background] Hernández Ávila M, Rivera Dommarco J, Shamah Levy T. Encuesta Nacional de Salud y Nutrición 2016. Resultados Nacionales. Cuernavaca, México: Instituto Nacional de Salud Pública (MX), 2016.
- [Background] Cueto Manzano AM, Cortés Sanabria L, Martínez Ramírez HR, et al. Enfermedad Renal Crónica Temprana: Prevención, diagnóstico y tratamiento. México: Médica Panamericana; 2013. pp. 250.
- [Background] Wolf G. New insights into the pathophysiology of diabetic nephropathy: from haemodynamics to molecular pathology. Eur J Clin Invest. 2004 Dec;34(12):785-96. doi: 10.1111/j.1365-2362.2004.01429.x. PMID 15606719
- [Background] Navarro JF, Milena FJ, Mora C, Leon C, Garcia J. Renal pro-inflammatory cytokine gene expression in diabetic nephropathy: effect of angiotensin-converting enzyme inhibition and pentoxifylline administration. Am J Nephrol. 2006;26(6):562-70. doi: 10.1159/000098004. Epub 2006 Dec 13. PMID 17167242
- [Background] Uruno A, Furusawa Y, Yagishita Y, Fukutomi T, Muramatsu H, Negishi T, Sugawara A, Kensler TW, Yamamoto M. The Keap1-Nrf2 system prevents onset of diabetes mellitus. Mol Cell Biol. 2013 Aug;33(15):2996-3010. doi: 10.1128/MCB.00225-13. Epub 2013 May 28. PMID 23716596
- [Background] Gómez García EF, Martínez Ramírez HR, Cortés Sanabria L, et al. Cambios y mejoras en la calidad de la dieta en pacientes con enfermedad renal crónica temprana. En: Conferencia dentro del marco del XLVII Congreso Nacional de Nefrología; 2013 Sep 4-12; Guadalajara, Jalisco. México.
- [Background] Balagopal P, George D, Patton N, Yarandi H, Roberts WL, Bayne E, Gidding S. Lifestyle-only intervention attenuates the inflammatory state associated with obesity: a randomized controlled study in adolescents. J Pediatr. 2005 Mar;146(3):342-8. doi: 10.1016/j.jpeds.2004.11.033. PMID 15756217
- [Background] Ruiz S, Pergola PE, Zager RA, Vaziri ND. Targeting the transcription factor Nrf2 to ameliorate oxidative stress and inflammation in chronic kidney disease. Kidney Int. 2013 Jun;83(6):1029-41. doi: 10.1038/ki.2012.439. Epub 2013 Jan 16. PMID 23325084
- [Background] Yoh K, Hirayama A, Ishizaki K, Yamada A, Takeuchi M, Yamagishi S, Morito N, Nakano T, Ojima M, Shimohata H, Itoh K, Takahashi S, Yamamoto M. Hyperglycemia induces oxidative and nitrosative stress and increases renal functional impairment in Nrf2-deficient mice. Genes Cells. 2008 Nov;13(11):1159-70. doi: 10.1111/j.1365-2443.2008.01234.x. PMID 19090810
- [Background] Choi BH, Kang KS, Kwak MK. Effect of redox modulating NRF2 activators on chronic kidney disease. Molecules. 2014 Aug 20;19(8):12727-59. doi: 10.3390/molecules190812727. PMID 25140450
- [Background] Atul A and Lakhwinder S. Pathogenesis of diabetic nephropathy and potential therapeutic effect of curcumin: A Review. Int J Pharm Bio Sci 2013;4:79-87.